CLINICAL TRIAL: NCT07397936
Title: Rebamipide Versus Diquafosol-Cyclosporine for Perioperative Dry Eye Disease in Cataract Surgery: A Randomized Trial
Brief Title: Rebamipide Versus Diquafosol and Cyclosporine for Perioperative Dry Eye in Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Dong Hui Lim, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRF-2021R1C1C1007795
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease (DED); Cataract
MeSH Terms: conditions — Dry Eye Syndromes; Cataract | interventions — rebamipide; Ophthalmic Solutions; diquafosol; Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group R (Experimental): Participants receive topical rebamipide 2% ophthalmic solution four times daily, initiated 1 month before cataract surgery and continued for 3 months postoperatively.
  Interventions: Drug: Rebamipide 2% ophthalmic solution
- Group DC (Active Comparator): Participants receive topical diquafosol 3% ophthalmic solution four times daily in combination with cyclosporine 0.05% ophthalmic solution twice daily, initiated 1 month before cataract surgery and continued for 3 months postoperatively.
  Interventions: Drug: Diquafosol 3% ophthalmic solution; Drug: Cyclosporine 0.05% ophthalmic solution

INTERVENTIONS:
Drug: Rebamipide 2% ophthalmic solution — Topical administration, four times daily
  Arms: Group R
Drug: Diquafosol 3% ophthalmic solution — Topical administration, four times daily
  Arms: Group DC
Drug: Cyclosporine 0.05% ophthalmic solution — Topical administration, two times daily
  Arms: Group DC

SUMMARY:
The goal of this clinical trial is to compare the efficacy of 2% rebamipide monotherapy versus a combination therapy of 3% diquafosol and 0.05% cyclosporine for the management of dry eye disease in patients undergoing cataract surgery. It will also evaluate the safety and ocular surface stability effects of these treatments during the perioperative period.

The main questions it aims to answer are:

Does rebamipide monotherapy maintain tear film breakup time (TBUT) and prevent corneal damage as effectively as the combination therapy after surgery? How do patient symptoms (OSDI scores) and inflammation markers (MMP-9) change with each treatment?

Researchers will compare the rebamipide group to the diquafosol-cyclosporine combination group to evaluate their effects on perioperative dry eye management.

Participants will:

Use the assigned study eye drops starting 1 month before their cataract surgery and continuing for 3 months after surgery.

Visit the clinic for eye examinations at baseline, the day of surgery, and at 1 week, 1 month, and 3 months postoperatively.

Undergo tests including tear film breakup time measurement, corneal staining, Schirmer's test, and tear MMP-9 level assessments.

DETAILED DESCRIPTION:
Dry eye disease (DED) is common in patients undergoing cataract surgery and may worsen during the perioperative period, leading to ocular discomfort and delayed visual recovery. Pharmacologic treatments targeting tear film instability and ocular surface inflammation are therefore important in perioperative management.

This prospective, randomized, parallel-group clinical trial compared two perioperative treatment strategies for DED in patients scheduled for cataract surgery. Eligible participants with pre-existing dry eye disease were randomized in a 1:1 ratio to receive either topical rebamipide 2% monotherapy or combination therapy with topical diquafosol 3% and cyclosporine 0.05%. Study medications were initiated 1 month prior to surgery and continued for 3 months postoperatively.

The primary outcome measure was the change in tear film breakup time (TBUT) during the early postoperative period. Secondary outcome measures included changes in corneal staining graded by the Oxford scale, patient-reported symptoms assessed by the Ocular Surface Disease Index (OSDI), tear secretion measured by Schirmer's test, and ocular surface inflammation evaluated using a tear matrix metalloproteinase-9 (MMP-9) point-of-care immunoassay.

Clinical assessments were performed at baseline, on the day of surgery, and at postoperative week 1, month 1, and month 3. Safety was evaluated by monitoring intraoperative and postoperative adverse events throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for cataract surgery
* Presence of dry eye disease, defined as an Ocular Surface Disease Index (OSDI) score ≥12 and at least one of the following:

  * Tear film breakup time (TBUT) ≤7 seconds
  * Oxford corneal staining grade ≥1
  * Schirmer's test value ≤10 mm/5 min
* Ability and willingness to comply with the study protocol and follow-up schedule
* Provision of written informed consent

Exclusion Criteria:

* Presence of ocular surface or ocular conditions that could affect dry eye status (e.g., active keratitis or ocular infection)
* Use of topical intraocular pressure-lowering medications
* History of ocular surgery other than cataract surgery in the study eye
* Any systemic or ocular condition judged by the investigator to interfere with study participation or outcome assessment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Tear Film Breakup Time (TBUT) | From baseline to postoperative week 1
  Change in tear film breakup time (TBUT) from baseline and during the early postoperative period following cataract surgery, comparing rebamipide monotherapy with diquafosol-cyclosporine combination therapy.

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Score | From baseline to 1 and 3 months postoperatively
  Change in patient-reported ocular symptoms assessed using the Ocular Surface Disease Index (OSDI) questionnaire, comparing rebamipide monotherapy with diquafosol-cyclosporine combination therapy.
Change in Corneal Staining Grade (Oxford Scale) | From baseline to postoperative week 1, and to 1 and 3 months postoperatively
  Change in corneal epithelial staining graded using the Oxford grading scale following fluorescein staining, comparing ocular surface stability between treatment groups.
Change in Schirmer's Test Value | From baseline to 1 and 3 months postoperatively
  Change in tear secretion measured by Schirmer's test without anesthesia, comparing tear production between rebamipide monotherapy and diquafosol-cyclosporine combination therapy.
Change in Tear Matrix Metalloproteinase-9 (MMP-9) Level | From baseline to 1 and 3 months postoperatively
  Change in tear matrix metalloproteinase-9 (MMP-9) levels assessed using a point-of-care immunoassay (InflammaDry), comparing ocular surface inflammation between treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The detailed study protocol and the data that support the findings of this study are available from the corresponding author upon reasonable request.